CLINICAL TRIAL: NCT01566019
Title: Molecular Screening Analysis Used as Decision Tool for Targeted Molecular Treatment
Brief Title: Molecular Screening for Cancer Treatment Optimization
Acronym: MOSCATO 02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-A00841-40; 2011/1755 (Other: CSET number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Solid Tumors (Any Localization)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with non curable metastatic cancer (Experimental)
  Interventions: Procedure: Tumoral biopsy

INTERVENTIONS:
Procedure: Tumoral biopsy — Every enrolled patient undergoes tumoral biopsy

SUMMARY:
The primary objective of the study is to use high throughput molecular analysis (CGH Array and sequencing) to treat patients with metastatic cancer with targeted therapeutics in order to improve the progression free survival compared to the previous treatment line.

The secondary objectives are to investigate clinical practical feasibility of such technics, to potentially improve the overall survival of patients and to describe molecular portrait of Phase 1 candidates.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors ; Stade IV ; Local relapse or metastatic ; Uncurable
* Age > 6 months
* PS 0/1 or Lansky play scale >= 70%
* Minimum one treatment line, no limit in the prior number of treatment line
* Evaluable or measurable disease

Exclusion Criteria:

* Life expectancy < 3 months
* Carcinomatous meningitis
* Symptomatic or progressive radiologic brain metastasis for non-CNS tumors
* Polynuclear neutrophil < 1 x 10^9/L
* Platelets < 100 x 10^9/L
* Hemoglobin < 90 g/L
* ALT/AST > 2.5 N
* bilirubin > 1.5 N
* Creatinine >1.5 N
* Calcemia > ULN
* Phosphate > ULN
* Coagulation anomaly non-indicated for biopsy

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2150 (Estimated)
Dates: Start 2011-10-28 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) using a targeted treatment selected by molecular profiling compared to the PFS for the most recent regimen | From date of start of targeted treatment oriented by MOSCATO until the date of first progression or date of death from any cause, whichever came first, assessed up to 1 year
  Progression according to RECIST criteria or clinical progression or death of any cause

SECONDARY OUTCOMES:
Number of patient who received a targeted treatment oriented by molecular profiling | From the start to the end of enrollment, up to 3 years
  Number of patient who received a targeted treatment oriented by molecular profiling
Progression free Survival, Overall Survival and Response Rate | Until progression, up to 1 year
  Comparison of Progression Free Survival, Overall Survival and Response Rate between patients with targeted treatment and others enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles SORIA, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Martin-Romano P, Colmet-Daage L, Morel D, Baldini C, Verlingue L, Bahleda R, Gazzah A, Champiat S, Varga A, Michot JM, Ngo-Camus M, Nicotra C, Marabelle A, Soria JC, Rouleau E, Lacroix L, Hollebecque A, Massard C, Postel-Vinay S. Epigenetic gene alterations in metastatic solid tumours: results from the prospective precision medicine MOSCATO and MATCH-R trials. Eur J Cancer. 2022 Sep;173:133-145. doi: 10.1016/j.ejca.2022.06.014. Epub 2022 Jul 21. PMID 35872509
- [Derived] Verlingue L, Hollebecque A, Lacroix L, Postel-Vinay S, Varga A, El Dakdouki Y, Baldini C, Balheda R, Gazzah A, Michot JM, Marabelle A, Mir O, Arnedos M, Rouleau E, Solary E, De Baere T, Angevin E, Armand JP, Michiels S, Andre F, Deutsch E, Scoazec JY, Soria JC, Massard C. Human epidermal receptor family inhibitors in patients with ERBB3 mutated cancers: Entering the back door. Eur J Cancer. 2018 Mar;92:1-10. doi: 10.1016/j.ejca.2017.12.020. Epub 2018 Feb 3. PMID 29413684
- [Derived] Verlingue L, Malka D, Allorant A, Massard C, Ferte C, Lacroix L, Rouleau E, Auger N, Ngo M, Nicotra C, De Baere T, Tselikas L, Ba B, Michiels S, Scoazec JY, Boige V, Ducreux M, Soria JC, Hollebecque A. Precision medicine for patients with advanced biliary tract cancers: An effective strategy within the prospective MOSCATO-01 trial. Eur J Cancer. 2017 Dec;87:122-130. doi: 10.1016/j.ejca.2017.10.013. Epub 2017 Nov 14. PMID 29145038
- [Derived] Jovelet C, Ileana E, Le Deley MC, Motte N, Rosellini S, Romero A, Lefebvre C, Pedrero M, Pata-Merci N, Droin N, Deloger M, Massard C, Hollebecque A, Ferte C, Boichard A, Postel-Vinay S, Ngo-Camus M, De Baere T, Vielh P, Scoazec JY, Vassal G, Eggermont A, Andre F, Soria JC, Lacroix L. Circulating Cell-Free Tumor DNA Analysis of 50 Genes by Next-Generation Sequencing in the Prospective MOSCATO Trial. Clin Cancer Res. 2016 Jun 15;22(12):2960-8. doi: 10.1158/1078-0432.CCR-15-2470. Epub 2016 Jan 12. PMID 26758560